CLINICAL TRIAL: NCT05637229
Title: A Serosurvey Study of Hand, Foot, and Mouth Disease in Healthy Children Aged 6 to 71 Months Old in Bandung and West Bandung District, Indonesia
Brief Title: A Serosurvey Study of Hand, Foot, and Mouth Disease in Indonesia
Status: Completed | Type: Observational
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-EV71-4101
Record Dates: First submitted 2022-11-08; First posted 2022-12-05 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Hand, Foot and Mouth Disease
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a sero-survey study of infants aged 6 months to 71 months in Bandung City and West Bandung District. As initial data to find out how many children have been exposed to human enterovirus type 71 (HEV-71) which causes Hand, foot, and mouth disease (HFMD).

DETAILED DESCRIPTION:
This study is a cross-sectional seroprevalence survey of EV-71, associated with HFMD, among children aged between 6 to 71 months in Bandung, sampled from urban and rural Primary Health Center in Bandung, Indonesia. This study was implemented by Department of Child Health Hasan Sadikin General Hospital/Medical Faculty Universitas Padjadjaran Bandung, West Java. Age-stratified sample of 600 children aged 6-71 months will be conducted from these sites. Samples testing includes routine blood counts, enzyme-linked immunosorbent assays (ELISAs) for enterovirus type 71 (EV71) IgG and ELISAs for other HFMD-associated enteroviruses.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to 71 months.
* The participant's parent/guardian receives an explanation and receives a Letter of Consent after the explanation (informed consent) and provided a documented informed consent by parents/legally accepted representative (LAR) participants prior to the study procedures.
* Domicile in Bandung and West Bandung District for at least 6 months.

Exclusion Criteria:

* Children with difficulty to withdraw the blood during blood collection
* Children with severe illness who require further treatment

Ages: 6 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population are children aged between 6 to 71 months in Bandung, sampled from urban and rural Primary Health Center in Bandung, Indonesia
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Seroprevalence of EV71 antibodies | Immediately after sampling
  Proportion of participants who are seropositive (IgG) for EV-71 and proportion of participants who are seropositive for EV-71 per predefined age-groups (6 - 35 months and 36 - 71 months)

SECONDARY OUTCOMES:
Proportion of abnormality result for Routine blood tests | Immediately after sampling
  Proportion of abnormality result for Routine blood tests (Red blood cells, white blood cells, platelets, haemoglobin, haematocrit).
seroprevalence of other HFMD-associated enteroviruses antibodies | Immediately after sampling
  Proportion of participants who are seropositive (IgG) for and other HFMD-associated enteroviruses and proportion of participants who are seropositive for and other HFMD-associated enteroviruses per predefined age-groups (6 - 35 months and 36 - 71 months)

CONTACTS AND LOCATIONS:
Overall Officials: Rodman Tarigan, Doctor, Principal Investigator — Hasan Sadikin Hospital/School of Medicine, Padjadjaran University, Bandung
Locations (2):
- Indonesia (2):
  - Garuda Health Center, Bandung
  - Padalarang Health Center, Bandung

REFERENCES:
- [Derived] Girsang RT, Rusmil K, Fadlyana E, Setiabudiawan B, Adrizain R, Mulyadi RP, Budiman A, Utami RK, Mardiah BZ, Dwi Putra MG, Fulendry FP, Nashsyah DT, Sukandar H. A serosurvey study of hand, foot and mouth disease in healthy children aged 6 to 71 months old in West Bandung and Bandung Region, Indonesia. BMC Infect Dis. 2025 Jan 27;25(1):124. doi: 10.1186/s12879-025-10453-0. PMID 39871167